CLINICAL TRIAL: NCT02915731
Title: Total Body Vitamin A Pool Size in Preschool Children Before and After Vitamin A Supplementation in an Impoverished South African Community Where Liver is Frequently Eaten and Children Exposed to Vitamin A Fortified Staple Foods
Brief Title: Total Body Vitamin A Before and After Vitamin A Supplementation in a Community Where Liver is Frequently Eaten
Status: Completed | Type: Observational
Sponsor: Medical Research Council, South Africa (Other)
Collaborators: International Atomic Energy Agency (Other Government); University of Wisconsin, Madison (Other)
Responsible Party: Principal Investigator, Lize van Stuijvenberg, Senior Specialist Scientist, Medical Research Council, South Africa
Other Study IDs: EC016-5/2015
Record Dates: First submitted 2016-08-30; First posted 2016-09-27 (Estimated); Last update posted 2016-09-27 (Estimated); Status verified 2016-09

CONDITIONS: Hypervitaminosis A
Keywords: Vitamin A stores; Stable isotope dilution; Multiple vitamin A interventions
MeSH Terms: conditions — Hypervitaminosis A

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Dietary Supplement: Vitamin A supplement — 200 000 IU vitamin A (once-off dose), given to participants as part of the national vitamin A supplementation program

SUMMARY:
This study will assess total body vitamin A pool size, as well as liver vitamin A stores, by means of stable isotope dilution in preschool children from a South African community where liver, an exceptionally rich source of vitamin A, is frequently eaten, and the children exposed to vitamin A fortified staple foods, as well as a vitamin A supplementation programme.

DETAILED DESCRIPTION:
Serum retinol, the most commonly used indicator to assess vitamin A status, is homeostatically controlled and, although it is able to detect deficiency, it does not necessarily reflect liver stores or measure excessive vitamin A intake. The stable isotope dilution method is able to measure total vitamin A body pool size over the vitamin A status continuum, including the sub-toxic range,and would add valuable information about the vitamin A status in a community where liver (an exceptionally rich source of vitamin A) is frequently eaten, and children also exposed to other vitamin A interventions. Total body vitamin A will be assessed before and 4 weeks after a high dose vitamin A supplement given to the children as part of the national vitamin A supplementation program. The confounding effect of infection/inflammation on the biomarkers of vitamin A status will also be examined, as well as how serum retinol and retinol binding protein relate to each other, and to vitamin A pool size.

ELIGIBILITY:
Inclusion Criteria:

* Living in the study area;
* Must not have received a vitamin A supplement in the preceding month

Exclusion Criteria:

* Severe anaemia (haemoglobin < 9 g/dL);
* Fever (body temperature > 38°C)

Ages: 36 Months to 60 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: 3-5 year-old children from a low socio-economic South African community where liver is frequently eaten
Sampling Method: Non-Probability Sample
Enrollment: 95 (Actual)
Dates: Start 2016-04; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Number of participants with total body vitamin A stores in the sub-toxic range as measured by stable isotope dilution using 13C-retinol as tracer | 4 weeks

SECONDARY OUTCOMES:
Number of participants with elevated inflammation markers, as measured by elevated C-reactive protein (CRP) and alpha-1-acid glycoprotein (AGP), and their confounding effect on serum retinol, retinol binding protein, and body vitamin A stores | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Martha E van Stuijvenberg, PhD, Principal Investigator — Medical Research Council, South Africa; Muhammad A Dhansay, FC Paed, Principal Investigator — Medical Research Council, South Africa
Locations (1):
- South African Medical Research Council, Cape Town, South Africa

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] van Stuijvenberg ME, Schoeman SE, Lombard CJ, Dhansay MA. Serum retinol in 1-6-year-old children from a low socio-economic South African community with a high intake of liver: implications for blanket vitamin A supplementation. Public Health Nutr. 2012 Apr;15(4):716-24. doi: 10.1017/S1368980011002126. Epub 2011 Aug 23. PMID 21859509
- [Background] Nel J, van Stuijvenberg ME, Schoeman SE, Dhansay MA, Lombard CJ, du Plessis LM. Liver intake in 24-59-month-old children from an impoverished South African community provides enough vitamin A to meet requirements. Public Health Nutr. 2014 Dec;17(12):2798-805. doi: 10.1017/S1368980013003212. Epub 2013 Nov 28. PMID 24476795
- [Background] Tanumihardjo SA. Usefulness of vitamin A isotope methods for status assessment: from deficiency through excess. Int J Vitam Nutr Res. 2014;84 Suppl 1:16-24. doi: 10.1024/0300-9831/a000182. PMID 25537102
- [Derived] Sheftel J, van Stuijvenberg ME, Dhansay MA, Suri DJ, Grahn M, Keuler NS, Binkley NC, Tanumihardjo SA. Chronic and acute hypervitaminosis A are associated with suboptimal anthropometric measurements in a cohort of South African preschool children. Am J Clin Nutr. 2022 Apr 1;115(4):1059-1068. doi: 10.1093/ajcn/nqab422. PMID 35030234
- [Derived] van Stuijvenberg ME, Dhansay MA, Nel J, Suri D, Grahn M, Davis CR, Tanumihardjo SA. South African preschool children habitually consuming sheep liver and exposed to vitamin A supplementation and fortification have hypervitaminotic A liver stores: a cohort study. Am J Clin Nutr. 2019 Jul 1;110(1):91-101. doi: 10.1093/ajcn/nqy382. PMID 31089689